CLINICAL TRIAL: NCT02799277
Title: A Multinomial Process Model of Moral Judgment
Acronym: PSY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2014-12-0010
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Testosterone; Placebos
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Testosterone (Experimental): 14mg testosterone will be administered intranasally in a 1milliliter aqueous solution
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): 1ml blank (containing no drug) aqueous solution will be administered intranasally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — Effect of testosterone on moral decision making
  Arms: Testosterone
Drug: Placebo — Effect of testosterone on moral decision making
  Arms: Placebo

SUMMARY:
The main goal of this project to investigate the psychological processes underlying moral judgments in social dilemmas. We will examine neuroendocrine determinants of moral judgment by investigating the effects of exogenous testosterone

DETAILED DESCRIPTION:
* Medical Screening Interview: Participants will be asked to answer several questions to identify potential medical and non-medical conditions that would preclude the self-administration of testosterone.
* First Saliva Sample: Participants will be asked provide a saliva sample after they completed the medical screening interview.
* Testosterone Self-Administration: Immediately following the first saliva collection, participants will self-administer spray puffs of either testosterone or placebo.
* Relaxation: Participants will be given the opportunity to relax for 30 minutes.
* Moral Dilemmas Judgments: Participants will be asked to read a set of 24 moral dilemmas that describe situations in which an actor has to make a decision on whether or not to engage in a particular action (e.g., sacrifice the well-being of one person to protect the well-being of several others). Participants will be asked to indicate whether they consider the described action acceptable or unacceptable.
* Demographics: Participants will be asked to indicate their gender, age, and ethnicity.
* Ear Temperature, heart rate, and blood pressure will be measured before drug administration, and again 20 minutes after drug administration. If temperature changes more than 2 degrees, heart rate changes more than 20bmp, or if blood pressure changes more than 20%, the experiment will be terminated and subjects will be escorted across the street to the University Emergency Room.

ELIGIBILITY:
Inclusion Criteria:

* must be currently enrolled at The University of Texas at Austin

Exclusion Criteria:

* not comfortable with the self-administration of testosterone for the purpose of our study less than 18 years old BMI less than 18 or above 27 suffer from any of the physical health conditions listed on the pre-screen questionnaire (I will not ask about mental health because our study is not about mental health) take any of the medications listed on the pre-screen questionnaire currently pregnant (females) irregular cycle in the past 6 months (females) smoke more than 5 cigarettes/day use cocaine more than once/month (**or should I exclude all those who use any drugs recreationally more than once/month?**) drink more than 10 alcoholic beverages/week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Moral Dilemma Judgments | 90 minutes
  Subjects will decide on whether or not to engage in a particular action (e.g., sacrifice the well-being of one person to protect the well-being of several others). Participants will be asked to indicate whether they consider the described action acceptable or unacceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Josephs, PhD, Principal Investigator — Professor
Locations (1):
- University of Texas at Austin Department of Psychology, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No